CLINICAL TRIAL: NCT02533960
Title: Registry of Acute Stroke Under Novel Oral Anticoagulants - Prime
Acronym: RASUNOA-Prime
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); Daiichi Sankyo (Industry); University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Prof. Roland Veltkamp, Principal Investigator, University Hospital Heidelberg
Other Study IDs: RASUNOA-Prime
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage; Oral Anticoagulation; Cardiovascular Diseases; Vascular Diseases
Keywords: Registry of Acute Stroke Under Novel Oral Anticoagulants
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Cardiovascular Diseases; Vascular Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NOAC: Ischemic stroke substudy: inclusion of 1000 patients under treatment with non-vitamin K antagonist oral anticoagulants (NOACs).
  Hemorrhagic stroke substudy: inclusion of 334 patients under treatment with non-vitamin K antagonist oral anticoagulants (NOACs).
  Interventions: Other: not applicable (observational study)
- VKA: Ischemic stroke substudy: inclusion of 1000 patients under treatment with vitamin K antagonists (VKA).
  Hemorrhagic stroke substudy: inclusion of 333 patients under treatment with vitamin K antagonists (VKA)
  Interventions: Other: not applicable (observational study)
- Without OAC: Ischemic stroke substudy: inclusion of 1000 patients without oral anticoagulation.
  Hemorrhagic stroke substudy: inclusion of 333 patients without oral anticoagulation.
  Interventions: Other: not applicable (observational study)

INTERVENTIONS:
Other: not applicable (observational study) — Observational study without study related intervention.

SUMMARY:
The Registry of Acute Stroke Under Novel Oral Anticoagulants-Prime (RASUNOA-Prime), an investigator-initiated study, is a German multicenter, prospective, observational registry. It is performed at about 50 certified stroke-units and supported by an unrestricted grant from different pharmaceutical companies to the Heidelberg University Hospital. RASUNOA-Prime is designed to assess the emergency management of acute ischemic and hemorrhagic stroke patients with atrial fibrillation (AF) under different anticoagulation schemes pre stroke: Non-vitamin K antagonist oral anticoagulants (NOAC), Vitamin K antagonists (VKA), and no anticoagulation.

DETAILED DESCRIPTION:
The main purpose of this observational cohort study is to assess routine emergency management of acute stroke patients with AF under different anticoagulation schemes before the index stroke.

The investigators will address the following aims and objectives:

1. Describing emergency management of stroke patients (IS and ICH) with AF in clinical routine including early diagnostic, therapeutic and preventive procedures and assessing variations in emergency management of patients with AF by anticoagulation schemes pre stroke.
2. Identifying variations in risk of early complications (e.g. symptomatic secondary intracerebral haemorrhage in ischemic stroke patients) with AF by different anticoagulation schemes pre stroke.
3. Determining factors influencing outcome of stroke patients with AF at three months and clarifying the potential influence of different anticoagulation schemes pre stroke.

The registry consists of 2 separate substudies that cover two different patient cohorts: ischemic stroke and intracerebral hemorrhage.

The study will collect information from prospectively enrolling Neurology departments with certified stroke units across Germany.

The principal investigator, Prof. Dr. med. Roland Veltkamp, is affiliated with Imperial College London, UK, and Heidelberg University Hospital, Germany.

ELIGIBILITY:
Ischemic stroke substudy:

Inclusion Criteria:

* Age >= 18 years
* Informed consent
* Acute ischemic stroke with either symptoms lasting ≥ 24h or evidence of infarction in brain imaging

  * Anticoagulation with NOAC
  * Anticoagulation with VKA
  * No anticoagulation
* Previous/present atrial fibrillation

Exclusion Criteria:

* No informed consent
* Symptom-onset > 24 h

Hemorrhagic stroke substudy:

Inclusion Criteria:

* Age >= 18 years
* Acute primary intracerebral hemorrhage
* - a) Anticoagulation with NOAC
* - b) Anticoagulation with VKA
* - c) No anticoagulation
* Previous/present atrial fibrillation

Exclusion Criteria:

* No informed consent
* Symptom-onset > 24 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients with atrial fibrillation (AF) under different anticoagulation schemes pre stroke [Non-vitamin K antagonists oral anticoagulants (NOAC, also referred to as novel or new oral anticoagulants), Vitamin K antagonists (VKA), and no oral anticoagulation. According to the type of stroke, patients will be enrolled in the ischemic or hemorrhagic stroke substudy.
  NOTE: As of July 2019, enrollment in the ischemic stroke substudy was terminated due to achievement of the targeted enrolling numbers.
  NOTE: As of April 2021, enrollment in the intracerebral hemorrhage substudy was terminated due to achievement of the targeted enrolling numbers.
Sampling Method: Probability Sample
Enrollment: 3832 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Primary hypothesis (ischemic stroke substudy) | Participants will be followed for the duration of hospital stay, an expected average of less than 2 weeks"
  Intracerebral hemorrhage complications (i.e. sICH, according to NINDS and SITS-MOST)
Primary hypothesis (hemorrhagic stroke substudy) | 24 hours
  Proportion of relevant secondary hematoma expansion on follow-up neuroimaging (hematoma expansion of >= 33% or 6 mL)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Veltkamp, Prof. Dr. med., Principal Investigator — Heidelberg University Hospital, Department of Neurology, Heidelberg, Germany; Department of Stroke Medicine, Imperial College London, London, United Kingdom.
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Haas K, Purrucker JC, Rizos T, Heuschmann PU, Veltkamp R. Rationale and design of the Registry of Acute Stroke Under Novel Oral Anticoagulants-prime (RASUNOA-prime). Eur Stroke J. 2019 Jun;4(2):181-188. doi: 10.1177/2396987318812644. Epub 2018 Dec 17. PMID 31259266